CLINICAL TRIAL: NCT04747015
Title: A Comparative Study Between Cervical Traction and Active Management of 3rd Stage of Labor in Prevention of Postpartum Hemorrhage After Vaginal Delivery
Brief Title: Cervical Traction vs. Active Management of 3rd Stage of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 61
Record Dates: First submitted 2020-07-10; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Watchful Waiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical traction (Active Comparator): sustained traction downward and posteriorly was applied to anterior and posterior lips of the cervix using ovum forceps for approximately 90 seconds. The traction should be adequate to allow the cervix to reach the vaginal introitus
  Interventions: Drug: Oxytocin; Procedure: cervical traction
- Active management (Active Comparator): administration of oxytocin 5 IU units IM (WHO GDG recommendations,2012) and waiting for signs of placental separation then controlled cord traction (CCT)to the umbilical cord while applying simultaneous counter-pressure to the uterus, through the abdomen(Brandt Andrews maneuver)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 10 IU I.V shot administered at the time of delivery of the anterior shoulder of the baby according to the WHO recommendation
  Other Names: Routine oxytocin
  Arms: Active management
Drug: Oxytocin — 5 IU units IM (WHO GDG recommendations,2012) and waiting for signs of placental separation then controlled cord traction (CCT)to the umbilical cord while applying simultaneous counter-pressure to the uterus, through the abdomen(Brandt Andrews maneuver)
  Other Names: Active management
Procedure: cervical traction — sustained traction downward and posteriorly was applied to anterior and posterior lips of the cervix using ovum forceps for approximately 90 seconds. The traction should be adequate to allow the cervix to reach the vaginal introitus. Meanwhile (CCT ) is avoided and watchful waiting for signs of placental separartion till 90 seconds end
  Other Names: Amr maneuver
  Arms: Cervical traction

SUMMARY:
306 patients will be divided randomly in to 2 GROUPS:

* control group: 153 patients will receive Oxytocin 10 IU I.V shot administered at the time of delivery of the anterior shoulder of the baby for both groups in prevention of postpartum haemorrhage,followed by active management of the third stage of labor by administration of oxytocin 5 IU units IM and waiting for signs of placental separation then controlled cord traction (CCT) to the umbilical cord while applying simultaneous counter-pressure to the uterus, through the abdomen(Brandt Andrews maneuver)
* study group:156 patients received Oxytocin 10 IU I.V shot at the time of delivery of the of the anterior shoulder of the baby according to the WHO recommendation .Then oxytocin is stopped and cervical traction (Amr maneuver )is applied.

In the maneuver,sustained traction downward and posteriorly was applied to anterior and posterior lips of the cervix using ovum forceps for approximately 90 seconds. The traction should be adequate to allow the cervix to reach the vaginal introitus. Meanwhile (CCT ) is avoided and watchful waiting for signs of placental separartion till 90 seconds end. Massage is not employed but the fundus is frequently palpaple to insure it doesnot become atonic and filled with blood from placenta separation. In cases whom placental separation did not occur within the 90 seconds, we removed the ovum forceps and waited for 30 min for the placental separation .

DETAILED DESCRIPTION:
The patients were divided randomly in to 2 GROUPS:

* control group: 153 patients received Oxytocin 10 IU I.V shot administered at the time of delivery of the anterior shoulder of the baby according to the WHO recommendation for both groups in prevention of postpartum haemorrhage,followed by active management of the third stage of labor by administration of oxytocin 5 IU units IM (WHO GDG recommendations,2012) and waiting for signs of placental separation then controlled cord traction (CCT)to the umbilical cord while applying simultaneous counter-pressure to the uterus, through the abdomen(Brandt Andrews maneuver)
* study group:156 patients received Oxytocin 10 IU I.V shot at the time of delivery of the of the anterior shoulder of the baby according to the WHO recommendation .Then oxytocin is stopped and cervical traction (Amr maneuver )is applied.

In the maneuver,sustained traction downward and posteriorly was applied to anterior and posterior lips of the cervix using ovum forceps for approximately 90 seconds. The traction should be adequate to allow the cervix to reach the vaginal introitus. Meanwhile (CCT ) is avoided and watchful waiting for signs of placental separartion till 90 seconds end. Massage is not employed but the fundus is frequently palpaple to insure it doesnot become atonic and filled with blood from placenta separation. In cases whom placental separation did not occur within the 90 seconds, we removed the ovum forceps and waited for 30 min for the placental separation .

ELIGIBILITY:
Inclusion Criteria:

singleton pregnancy full term pregnancy ( gestational age 37 - 42 weeks).

Exclusion Criteria:

* twin pregnancy, preterm labor <36 weeks, fetal macrosomia, any case with bleeding tendency e.g: haemorrhagic diseases and cases with risk of postpartum haemorrhage as: Peripartun hemorrhage ( placenta previa or placental abruption), anemia or hypertension

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 306 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
occurrence of postpartum hemorrhage | 24 hours after delivery
  blood loss more than 500 ml

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided